CLINICAL TRIAL: NCT00848523
Title: Phase II Trial of LBH589 (Panobinostat) in Adult Patients With Recurrent Malignant Gliomas
Brief Title: Study of LBH589 (Panobinostat) to Treat Malignant Brain Tumors
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: insufficient accrual
Sponsor: Neurological Surgery, P.C. (Other)
Responsible Party: J. Paul Duic, MD, Long Island Brain Tumor Center at Neurological Surgery, PC
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: LIBTC-2008-1
Record Dates: First submitted 2009-02-19; First posted 2009-02-20 (Estimated); Last update posted 2010-07-16 (Estimated); Status verified 2009-09

CONDITIONS: Recurrent Malignant Gliomas
Keywords: LBH859; Panobinostat; GBM; Glioma; Glioblastoma; Astrocytoma; oligodendroglioma; oligoastrocytoma; gliosarcoma; anaplastic
MeSH Terms: conditions — Glioma; Glioblastoma; Astrocytoma; Oligodendroglioma; Gliosarcoma | interventions — Panobinostat

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Panobinostat — 30 mg, three times a week, patients will continue with treatment until they experience unacceptable toxicity that precludes further treatment, disease progression, and/or at the discretion of the investigator.
  Other Names: LBH589

SUMMARY:
The drug LBH589 (panobinostat) is an experimental (investigational) drug that is being tested for recurrent (returning) malignant gliomas. An investigational drug is one that has not been approved by the U.S. Food and Drug Administration (FDA). It belongs to a new class of drugs called "histone deacetylase inhibitors." Histones are proteins located in the nucleus of cells that bind to DNA, the chemical that makes up genes. These proteins help control which genes are turned "on" and "off." Studies have shown that drugs like panobinostat (LBH589) may lead to tumor cell death.

DETAILED DESCRIPTION:
The prognosis for recurrent malignant gliomas remains dismal despite advances in neurological surgery, radiation oncology and chemotherapy. Median overall survival remains a mere 14.6 months and 2 yr survival 25% (Stupp et al.) Novel treatments are clearly needed for recurrent gliomas.

Preclinical data suggests that histone deacetylase inhibition may be an effective treatment for recurrent malignant gliomas.

In 1999, in the Proceedings of the National Academy of Sciences, Saito reported that MS-27-275, a benzamide derivative and inhibitor of histone deacetylase, inhibited the growth of several different human tumor cell lines.

The drug you are being asked to take is called LBH589 or panobinostat. It belongs to a new class of drugs called "histone deacetylase inhibitors." Histones are proteins located in the nucleus of cells that bind to DNA, the chemical that makes up genes. These proteins help control which genes are turned "on" and "off". Studies have shown that drugs like panobinostat (LBH589) may lead to tumor cell death.

Before starting on-study, we will require that some standard blood tests be done. You may have other tests done as well.

LBH589 (panobinostat) is a drug that you will take three times weekly by mouth on Monday, Wednesday and Friday. You will take the capsules with an 8 ounce glass of water (not grapefruit or orange juice) on an empty stomach at least 2 hours after meals and 2 hours before next meal. Cycles are twenty eight (28) days long.

The study drug may affect your heart rhythm. Therefore, we will closely monitor your heart by doing an electrocardiogram (ECG) while you are taking the study drug. On the first day that you start taking the drug, we will record your ECG at several different time points: three ECG's at 5 minute intervals before you take your first dose and then again at 2 hours, 4-6 hours and 24-32 hours after you take your first dose. On days 5 and 19 of the first cycle (the first twenty eight days) we will also obtain (3) more ECG's: one before you take your daily dose and then two more at 2 hours and 4-6 hours after taking the medication.

On future cycles (cycle 2 and thereafter) we will obtain single ECG's on days # 5 and 22 if there had been no prior abnormal readings.

You will return to clinic for follow-up examination midway through the first cycle and then again upon completion of the first cycle and each following cycle.

Follow-up blood tests will be obtained at the end of the first, second and fourth weeks of the first cycle and then at the end of each following cycle.

Follow-up MRI (or CAT) scans will be obtained according to standard of care after each second cycle unless medically indicated at other time points.

Other scans, such as PET scans, may be obtained if medically indicated as per standard of care.

ELIGIBILITY:
Inclusion Criteria:

* Recurrent malignant glioma with radiographic progression
* No more than three prior therapies.
* Male or female patients >=18 years old
* KPS >=60.
* Ability to provide written informed consent or consent obtained from responsible healthcare proxy.
* Contrast-enhanced MRI within 2 weeks of enrollment.
* Life expectancy >= 8 weeks
* Neutrophils >1500/mm3
* Platelets > 100,000/mm3L
* Hemoglobin >=9 g/dL
* AST/SGOT and ALT/SGPT <= 2.5 x upper limit of normal (ULN) or < 5.0 x ULN if the transaminase elevation is due to disease involvement
* Serum bilirubin <= 1.5 x ULN
* Serum creatinine <= 1.5 x ULN or 24-hour creatinine clearance >= 50 ml/min
* Total serum calcium or ionized calcium WNL
* Serum potassium WNL
* Serum sodium WNL
* Serum albumin >= LLN or 3g/dl
* Elevated Alkaline Phosphatase due to bone metastasis can be enrolled
* Baseline MUGA or ECHO must demonstrate LVEF >= the LLN
* TSH and free T4 WNL (patients may be on thyroid hormone replacement)
* Women of childbearing potential (WOCBP) must have a negative serum pregnancy test within 7 days of the first administration of study treatment and must be willing to use two methods of contraception one of them being a barrier method during the study and for 3 months after last study drug administration.
* No concurrent antitumor therapy.
* No enzyme-inducing antiepileptic drugs.
* No significant comorbidities
* Patients must have recovered from toxic effects of prior therapy.

Exclusion criteria

* Prior HDAC, DAC, HSP90 inhibitors or valproic acid for the treatment of cancer
* Valproic acid for any medical condition during the study or within 5 days prior to first LBH589 treatment
* Impaired cardiac function including:
* Screening ECG with a QTc > 450 msec
* Congenital long QT syndrome
* History of sustained ventricular tachycardia
* History of ventricular fibrillation or torsades de pointes
* Bradycardia < 50 beats per minute. Patients with a pacemaker and heart rate > = 50 beats per minute are eligible.
* Myocardial infarction or unstable angina within 6 months
* Congestive heart failure (NYHA class III or IV)
* RBBB and LAH (bifascicular block)
* Uncontrolled hypertension
* Concomitant use of drugs with a risk of causing torsades de pointes Concomitant use of CYP3A4 inhibitors
* Patients with unresolved diarrhea
* Impairment of gastrointestinal (GI) function or GI disease that may significantly alter absorption of LBH589
* Concurrent severe and/or uncontrolled medical conditions
* Chemotherapy, any investigational drug or major surgery < 4 weeks prior to starting study drug or have not recovered from side effects of such therapy.
* Concomitant use of any anti-cancer therapy or radiation therapy.
* Women who are pregnant or breast feeding or women of childbearing potential (WOCBP) not willing to use a double barrier method of contraception during the study and 3 months after the end of treatment. One of these methods of contraception must be a barrier method.
* Male patients whose sexual partners are WOCBP not using a double method of contraception during the study and 3 months after the end of treatment. One of these methods must be a condom
* History of another primary malignancy within 5 years other than curatively treated CIS of the cervix, or basal or squamous cell carcinoma of the skin
* Known human immunodeficiency virus (HIV) or hepatitis C positivity
* Significant history of non-compliance to medical regimens or inability to grant a reliable informed consent
* More than three prior therapies
* Hepatic or renal diseases or any diseases that will obscure toxicity or alter drug metabolism
* Known active malignancies
* Active infection requiring iv antibiotics
* Systemic anticoagulants
* Enzyme-inducing antiepileptic drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2008-11; Primary Completion 2009-04 (Estimated); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
To generate preliminary data of anti-tumor efficacy of LBH589 in adults with recurrent malignant gliomas. | 12 months

SECONDARY OUTCOMES:
To determine primary efficacy endpoint PFS-6 | 6 months
To determine objective response (CR + PR) Rate | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: J. Paul Duic, MD, Principal Investigator — Long Island Brain Tumor Center at Neurological Surgery PC / Long Island Neuro-Oncology Associates; Jai Grewal, MD, Principal Investigator — Long Island Brain Tumor Center at Neurological Surgery PC/ Long Island Neuro-oncology Associates
Locations (2):
- United States (2):
  - Long Island Brain Tumor Center at Neurological Surgery PC / Long Island Neuro-Oncology Associates, Commack, New York
  - Long Island Brain Tumor Center at Neurological Surgery PC / Long Island Neuro-Oncology Associates, Great Neck, New York